CLINICAL TRIAL: NCT06306625
Title: REmote Ischemic COnditioning in Out-of-Hospital Cardiac Arrest: The RECO-OHCA Study
Brief Title: REmote COnditioning in Out-of-Hospital Cardiac Arrest
Acronym: RECO-OHCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL21_0001; 2023-A01315-40 (Other: ID-RCB)
Record Dates: First submitted 2024-01-23; First posted 2024-03-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Out-of-hospital cardiac arrest; remote conditioning; ischemic conditioning; ischemia-reperfusion; intensive care unit
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic conditioning (Experimental): A brachial cuff is positioned around one arm of the patient. Remote ischemic conditioning consists of alternating inflations and deflations of the brachial cuff. Four cycles of ischemic conditioning (5-min brachial cuff inflation at 200 millimetres of mercury (mmHg) followed by 5-min cuff deflation) are started as soon as possible after inclusion. The intervention is repeated 12 and 24 hours after inclusion.
  Interventions: Device: Remote ischemic conditioning
- Control group (Other): A brachial cuff is positioned around one arm of the patient. Neither inflation nor deflation is performed.
  Interventions: Device: No remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — A brachial cuff is positioned around one arm of the patient. Remote ischemic conditioning consists of four cycles of a 5-min brachial cuff inflation at 200 mmHg followed by a 5-min of cuff deflation, and is started as soon as possible after randomization. The intervention is repeated 12 and 24 hours after inclusion.
  Arms: Remote ischemic conditioning
Device: No remote ischemic conditioning — A brachial cuff is positioned around the arm of the patient and no inflation or deflation is performed.
  Arms: Control group

SUMMARY:
Out-of-Hospital Cardiac Arrest remains a major public health problem, resulting in high mortality largely related to multiple organ failure and poor neurological outcomes due to brain anoxia. The pathophysiology of organ dysfunction after resuscitated out-of-hospital cardiac arrest involves ischemia-reperfusion processes. Remote ischemic conditioning is a therapeutic strategy used to protect organs against the detrimental effects of ischemia-reperfusion injury.

The objective of the present trial is to determine whether remote ischemic conditioning performed early after out-of-hospital cardiac arrest can decrease mortality, or multiple organ failure and/or severe neurological failure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* Out-of-hospital cardiac arrest, whatever the initial cardiac rhythm (shockable or non-shockable) or the duration of no-flow and low-flow,
* Presence of a witness who may or may not have started cardiopulmonary resuscitation, or patient seen alive in the 30 minutes prior to the cardiac arrest,
* Hospitalisation in critical care (intensive care unit or cardiac intensive care unit) for less than 3 hours,
* Informed consent obtained from a close relative (exceptionally from the patient himself if his condition permits) or, failing this, use of the emergency procedure by the investigator.

Exclusion Criteria:

* Traumatic cardiac arrest
* Patient on extracorporeal circulatory assistance
* Cardiac arrest for which continuation of resuscitation does not appear justified (unavoidable death, terminal stage of an irreversible disease, etc.)
* Contraindication of the use of brachial cuff on both arms (arteriovenous fistula, lymphoedema or severe peripheral vascular pathology, unstable humeral fracture, continuous infusion into an upper limb vein of an essential drug such as a catecholamine, radial arterial catheter for continuous invasive measurement of blood pressure)
* Pregnant, parturient, or breast-feeding women
* Patients deprived of their liberty by a judicial or administrative decision,
* Patients under legal protection (guardianship, curatorship),
* Patient not affiliated to a social security scheme or beneficiary of a similar scheme,
* Previous inclusion in the study,
* Subject participating in other interventional research that may interfere with the present study according to the investigator's judgement or that includes an exclusion period still in progress at inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
All cause of death | 72 hours after hospital admission
  All-cause death will be assessed 72 hours after hospital admission.
Multiple organ failure | 72 hours after hospital admission
  Multiple organ failure is defined by a SOFA (Sepsis-related Organ Failure Assessment) score, censored for the neurological component, greater than or equal to 5.
Severe neurological failure | 72 hours after hospital admission
  Severe neurological failure is defined by a motor component of the Glasgow Coma Score less than or equal to 3, without confounding factors (hypothermia less than or equal to 35.0°C, and/or sedation/analgesia/curarization).
  The glasgow coma score ranges from 3 to 15 and is broken down into its three parameters: eye opening, verbal response and motor response.
  The higher the score, the better the patient's recovery.

SECONDARY OUTCOMES:
Sepsis-related Organ Failure Assessment (SOFA) score | 24 hours after hospital admission
  The SOFA score ranges from 0 to 24 (higher scores indicate more severe organ failure), with 0 to 4 points assigned for each of 6 organ dysfunctions (ie, central nervous system, cardiovascular, respiratory, renal, coagulation, and liver).
Sepsis-related Organ Failure Assessment (SOFA) score | 48 hours after hospital admission
  The SOFA score ranges from 0 to 24 (higher scores indicate more severe organ failure), with 0 to 4 points assigned for each of 6 organ dysfunctions (ie, central nervous system, cardiovascular, respiratory, renal, coagulation, and liver).
Sepsis-related Organ Failure Assessment (SOFA) score | 72 hours after hospital admission
  The SOFA score ranges from 0 to 24 (higher scores indicate more severe organ failure), with 0 to 4 points assigned for each of 6 organ dysfunctions (ie, central nervous system, cardiovascular, respiratory, renal, coagulation, and liver).
Sepsis-related Organ Failure Assessment (SOFA) score after exclusion of the neurological sub-score | 24 hours after hospital admission
Sepsis-related Organ Failure Assessment (SOFA) score after exclusion of the neurological sub-score | 48 hours after hospital admission
Sepsis-related Organ Failure Assessment (SOFA) score after exclusion of the neurological sub-score | 72 hours after hospital admission
Sepsis-related Organ Failure Assessment (SOFA) sub-scores for each organ dysfunction | 24 hours after hospital admission
  Average SOFA sub-scores for each organ failure scored from 0 to 4 points
Sepsis-related Organ Failure Assessment (SOFA) sub-scores for each organ dysfunction | 48 hours after hospital admission
  Average SOFA sub-scores for each organ failure scored from 0 to 4 points
Sepsis-related Organ Failure Assessment (SOFA) sub-scores for each organ dysfunction | 72 hours after hospital admission
  Average SOFA sub-scores for each organ failure scored from 0 to 4 points
Mean Sepsis-related Organ Failure Assessment (SOFA) score | From hospital admission to 72 hours (or from hospital admission to death if it occurs before 72 hours)
Mean Sepsis-related Organ Failure Assessment (SOFA) score after exclusion of the neurological sub-score | From hospital admission to 72 hours (or from hospital admission to death if it occurs before 72 hours)
Variations of the Sepsis-related Organ Failure Assessment (SOFA) score (delta-SOFA) | Between hospital admission to 24 hours, admission to 48 hours and admission to 72 hours
Variations of the Sepsis-related Organ Failure Assessment (SOFA) score (delta-SOFA) after exclusion of the neurological sub-score | Between hospital admission to 24 hours, admission to 48 hours and admission to 72 hours
Serum level of neuron-specific enolase (NSE) | Between 48 and 72 hours after hospital admission
Cerebral Performance Categories (CPC) scale | Day 90
  The neurological performance is assessed using the cerebral performance categories (CPC) scale, which ranges from 1 to 5 (with 1 representing good cerebral performance or minor disability, 2 moderate disability, 3 severe disability, 4 coma or vegetative state, and 5 brain death or dead).
All-cause mortality | From date of randomization until day 90 after hospital admission

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Hôpital Louis Pradel, Bron
  - Hôpital Gabriel Montpied, CHU de Clermont Ferrand, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand, Clermont-Ferrand
  - Hôpital F Mitterrand, CHU de Dijon, Dijon
  - Hôpital Albert Michallon, CHU de Grenoble, La Tronche
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Saint-Joseph Saint-Luc, Lyon
  - Hôpital de la Timone, CHU de Marseille, Marseille
  - Hôpital lapeyronie, CHU de Montpellier, Montpellier
  - Hôpital Universitaire Carémeau, Nîmes
  - Hôpital Lariboisière, APHP, Réanimation Médicale et Toxicologique, Paris
  - Hôpital Lyon-Sud, Pierre-Bénite
  - Hôpital Nord, CHU de St Etienne, Saint-Priest-en-Jarez
  - Hôpital Nord-Ouest, Villefranche-sur-Saône